

**Project Title:** EDUCAT: An Assistive Powered Wheelchair. Stage 2. Powered Wheelchair User Evaluation of an Obstacle Alerting System.

NCT Number: NCT05292690

**Document Date: 29/06/2020** 



IRAS ID: 257062

Site name:

Participant Identification Number for this trial:

Title of Project: EDUCAT An Assistive Powered Wheelchair - Stage 2: User Evaluation of an Obstacle Alerting System

## **PARTICIPANT CONSENT FORM**

Please initial each box

| ( | . I confirm that I have read and understood the participant information sheet dated (version) for the above study. I have had the opportunity to consider the information, ask questions and have had these answered satisfactorily. | | | | |
|---|---|---|---|---|---|
| | 2. I understand my participation is voluntary and I am free to withdraw at any time without giving any reason, without my medical care or legal rights being affected. | | | | |
| | 3. I understand that even if I withdraw from the study, the data collected from me up to that point will be used in analysing the results of the study. | | | | |
| looked at but where it is | 4. I understand that relevant sections of my medical and research records may be looked at by authorised personnel from [site name] and regulatory authorities where it is relevant to my taking part in this research. I give permission for these individuals to have access to my records. | | | | |
| | 5. I understand that <b>anonymised</b> data collected during the study may be looked at by individuals from the EDUCAT project partners for analysis purposes. | | | | |
| | • | - | • • | for up to 10 years for projects in the future? | |
| be used to | 7. I understand and agree that the GPS system in the Obstacle Alerting System can be used to identify my location when outdoors. This information will only be used to help correlate my joystick movements with the nature of that location. | | | | |
| 8. I agree to ta | ake part in the | above research stu | dy. | | |
| Name of PWC User | | Date | | Signature | |
| Name of Person taking consent | | Date | | Signature | _ |



| Insert local site contact details:- |
|--------------------------------------------------------------------|
| Name of PI and/or researcher |
| Contact details: |
| NB. Original consent form for site file, one copy for participant. |